CLINICAL TRIAL: NCT00042913
Title: A Phase 2 Open Label, Randomized, Dose And Schedule Finding, Clinical Trial Of Immunotherapy With AMG 412 In Subjects With Diffuse Large B-Cell Non-Hodgkin's Lymphoma
Brief Title: Epratuzumab in Treating Patients With Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000069484; UCLA-0201056; AMGEN-AMG-412-159; NCI-G02-2094
Record Dates: First submitted 2002-08-05; First posted 2003-01-27 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2003-09

CONDITIONS: Lymphoma
Keywords: recurrent adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — epratuzumab

INTERVENTIONS:
Biological: epratuzumab

SUMMARY:
RATIONALE: Monoclonal antibodies such as epratuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Randomized phase II trial to study the effectiveness of epratuzumab in treating patients who have non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate of patients with diffuse large B-cell non-Hodgkin's lymphoma treated with epratuzumab.
* Determine the toxicity of this drug in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive low-dose epratuzumab IV over 1 hour once weekly for 4 weeks.
* Arm II: Patients receive low-dose epratuzumab IV over 1 hour once weekly for 8 weeks.
* Arm III: Patients receive high-dose epratuzumab IV over 1 hour once weekly for 4 weeks.

Patients are followed every 3 months for 2 years and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 150 patients (50 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diffuse large B-cell non-Hodgkin's lymphoma (NHL)

  * Relapsed or refractory after at least 1 regimen of standard therapy

    * Prior therapy may include high-dose chemotherapy with autologous stem cell transplantation (ASCT) or immunotherapy
* Bidimensionally measurable disease

  * At least 1 lesion at least 1.5 cm by CT scan
* No primary or secondary CNS lymphoma
* No HIV-related lymphoma
* No known or suspected transformed lymphoma (prior or concurrent)
* No bulky disease (i.e., any single mass greater than 10.0 cm)
* No pleural effusion with positive cytology for lymphoma
* Most recent pathology specimen available for collection
* No rapid disease progression or symptoms that indicate disease progression requiring rapid intervention within the past 2 weeks (e.g., severe shortness of breath, severe pain, or gastrointestinal or genitourinary obstruction)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 4 months

Hematopoietic

* Absolute neutrophil count at least 1,000/mm3
* Platelet count at least 50,000/mm3 (transfusion independent)
* Hemoglobin at least 9.0 g/dL

Hepatic

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* AST and ALT less than 5 times ULN
* Hepatitis B surface antigen negative
* Hepatitis C negative

Renal

* Creatinine no greater than 2 times ULN

Other

* HIV negative
* No other primary malignancy within the past 3 years except squamous cell or basal cell skin cancer, carcinoma in situ of the cervix, or stage I prostate cancer
* No other serious nonmalignant condition that would preclude study
* No serious infection
* No known human antichimeric antibodies or human antihuman antibody positivity
* No type 1 hypersensitivity or anaphylactic reactions to murine proteins
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 6 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* At least 4 weeks since prior immunotherapy (unless clearly progressing)
* At least 12 weeks since prior ASCT

Chemotherapy

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (unless clearly progressing)

Endocrine therapy

* Not specified

Radiotherapy

* No prior radioimmunotherapy

Surgery

* At least 4 weeks since prior major surgery (unless patient has fully recovered)

Other

* At least 30 days since prior enrollment in clinical trials involving investigational devices or drugs
* No concurrent enrollment in other clinical trials involving investigational devices or drugs
* No concurrent investigational agents for disease other than NHL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-05

CONTACTS AND LOCATIONS:
Overall Officials: Christos E. Emmanouilides, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States